CLINICAL TRIAL: NCT00822016
Title: INST 0701C: An Observational Outcomes Protocol of Standard Practice of Best Supportive Care With or Without Surgery, Chemotherapy or Radiotherapy in Patients With Carcinoma of the Lung
Brief Title: Observational Study of Best Supportive Care With or Without Surgery, Chemo or Radiotherapy in Pts With Carcinoma of Lung
Status: Terminated | Type: Observational
Why Stopped: PI left institution. Insufficient enrollment for analysis.
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0701C
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: Best Supportive Care; Protocol of Standard Practice; Carcinoma of the Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to establish a listing (database) of patients diagnosed with lung cancer and treated with best supportive care and standard and investigational chemotherapy regimens, surgery, and radiation therapy at the UNM CRTC and other NMCCA sites. The information will be used to determine the results of various treatments for lung cancer subjects and to find where improvements can be made in safety, effectiveness, supportive care, treatment that eases tumors without curing them, treatments that cure tumors, prevention, and follow-up efforts. The database information will be compared to clinical trial data published in peer-reviewed journals and SEER outcome data. Patients will be acquired both before and after they are treated for lung cancer.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Those who are eligible for this treatment protocol will consist of:

  1. Patients with histologically diagnosed lung cancer.
  2. Patients receiving therapy should have an ECOG/Zubrod/SWOG performance status of <3 at the time of the initiation of therapy.
  3. All newly diagnosed patients referred to an NMCC Alliance site will be eligible, as will patients with recurrent disease that are now referred to an NMCCA for their next therapy (such as those who move from out of state, or are referred for protocol therapy), though efforts will be made to obtain records of prior therapy administered elsewhere).

Exclusion Criteria:

* Patients not falling under any of the above criteria are not eligible for the study.
* Withdrawal of the informed consent at any point in the study excludes patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with lung cancer and treated with best supportive care and standard and investigational chemotherapy regimens, surgery, and radiation therapy at the UNM CRTC and other NMCCA sites.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To document the progression-free survival, rate of response, median duration of response, & median overall survivals, of subjects receiving best supportive care with or without standard surgery, chemotherapy and/or radiation therapy for lung cancer | 3-6 months

SECONDARY OUTCOMES:
To document the incidence and severity of toxicities, and reversibility of toxicities of subjects as a function of the treatments rendered. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennie Jones, M.D., Principal Investigator — University of New Mexico Cancer Center
Locations (2):
- United States (2):
  - University of New Mexico Cancer Center @ Lovelace Medical Center, Albuquerque, New Mexico
  - Universtiy of New Mexico Cancer Center, Albuquerque, New Mexico